CLINICAL TRIAL: NCT01765829
Title: Randomized Multicentric Open-label Phase III Clinical Trial to Evaluate the Efficacy of Continual Treatment Versus Discontinuation Based in the Presence of Prodromes in a First Episode of Non-affective Psychosis.
Brief Title: Clinical Trial to Evaluate the Efficacy of Treatment vs Discontinuation in a First Episode of Non-affective Psychosis
Acronym: NONSTOP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NONSTOP
Record Dates: First submitted 2013-01-03; First posted 2013-01-10 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Psychosis Nos/Other
Keywords: Non Affective Psychosis; First episode; Discontinuation scheme
MeSH Terms: interventions — Aripiprazole; Olanzapine; Clopenthixol; clothiapine; Flupenthixol; Risperidone; Sulpiride; Trifluoperazine; Haloperidol; Quetiapine Fumarate; Paliperidone Palmitate; Chlorpromazine; pipothiazine; periciazine; Clozapine; Pimozide; Perphenazine; sertindole; Methotrimeprazine; Amisulpride; asenapine; Tiapride Hydrochloride; Droperidol; ziprasidone; Antipsychotic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antipsychotic treatment (Active Comparator): Antipsychotic treatment according to common clinical practice
  Drugs: Aripiprazole, Olanzapine, Zuclopenthixol, Clotiapine, Flupentixol, Risperidone, Sulpiride, Trifluoperazine, Haloperidol, Quetiapine, Paliperidone, Chlorpromazine, Pipotiazine, Flufenazine, Periciazine, Clozapine, Pimozide, Perfenazine, Sertindole, Levomepromazine, Amisulpride, Asenapine, Tiapride, Droperidol, Ziprasidone.
  Interventions: Drug: Antipsychotic treatment
- Discontinuation antipsychotic treatment (Experimental): Dose reduction of antipsychotic treatment (25% every 4 weeks).
  Interventions: Drug: Discontinuation antipsychotic treatment

INTERVENTIONS:
Drug: Discontinuation antipsychotic treatment — Dose reduction until withdrawal
  Other Names: Aripiprazole; Olanzapine; Zuclopenthixol; Clotiapine; Flupentixol; Risperidone; Sulpiride; Trifluoperazine; Haloperidol; Quetiapine; Paliperidone; Chlorpromazine; Pipotiazine; Flufenazine; Periciazine; Clozapine; Pimozide; Perfenazine; Sertindole; Levomepromazine; Amisulpride; Asenapine; Tiapride; Droperidol; Ziprasidone
  Arms: Discontinuation antipsychotic treatment
Drug: Antipsychotic treatment — Antipsychotic treatment is not modify during the study, it is administered according to common clinical practice
  Other Names: Antipsychotic drugs
  Arms: Antipsychotic treatment

SUMMARY:
The purpose of this study is to assess if patients who continue with antipsychotic treatment for 12 or more months show the same risk of relapse (measured by PANSS) that patients with the same medical condition who have followed a discontinuation treatment scheme based in the presence of prodromes.

The candidates should accomplish the following criteria: first episode of non-affective psychosis who have followed antipsychotic treatment for 12 months and who have already shown remission criteria.

DETAILED DESCRIPTION:
Randomized, open label, multicenter, phase III clinical trial. Number of subjects: 104. Age range: 18 - 55 years of both sex.

Timepoints for evaluation: Every two weeks, during the first six months after initiation of treatment discontinuation/continuation. Every four weeks during the remaining six months, to complete a total follow-up scheme of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult age from 18 to 55 years old
* Non-affective psychosis diagnosis (schizophrenia, schizoaffective, schizophreniform disorders, acute psychosis, other psychosis according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV).
* Antipsychotic treatment for 12 months since clinical stabilization. Clinical stabilization is defined in case of admission by medical discharge (not including voluntary discharge). In case of voluntary discharge or no admission to hospital, clinical stabilization can be defined by the psychiatrist according to medical history and the information provided by the family.
* No changes in the antipsychotic doses in the last 4 months.
* No suicide attempts in the last 12 months.
* Patient who shows remission criteria.
* Signed informed consent form.

Exclusion Criteria:

* Patient who is not fluent in Spanish language
* Patient who takes mood stabilizers (Lithium, antiepileptic drugs...)
* Dependency on alcohol or other substances of abuse (cannabis, cocaine...)
* History of brain injury with loss of consciousness for more than 1 hour, stroke or other central nervous system disorders.
* Intelligence testing (IQ) less than 70.
* Suicide attempt from stabilization.
* Pregnancy or planning to become pregnant during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Risk of relapse | 12 months
  The purpose of this study is to assess if patients who continue with antipsychotic treatment for 12 or more months show the same risk of relapse (measured by PANSS) that patients with the same medical condition who have followed a discontinuation treatment scheme based in the presence of prodromes.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ruiz Veguilla, MD, PhD, Study Chair — Virgen del Rocío Hospital
Locations (17):
- Spain (17):
  - Hospital de Basurto, Bilbao, Bilbao
  - Mental Health Unit Villamartín, Villamartín, Cádiz
  - Mental Health Unit Baza, Baza, Granada
  - Mental Health Unit Motril, Motril, Granada
  - Mental Health Unit Andújar, Andújar, Jaén
  - Mental Health Unit Martos, Martos, Jaén
  - Mental Health Unit Miraflores, Alcobendas, Madrid
  - Mental Health Unit Tetuán, Madrid, Madrid
  - Lafora Hospital, Madrid, Madrid
  - Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Mental Health Unit Valle del Guadalhorce, Cártama, Málaga
  - Mental Health Unit Las Lagunas, Fuengiróla, Málaga
  - Hospital Carlos Haya, Málaga, Málaga
  - Fundación Argibide, Pamplona, Navarre
  - Hospital El Tomillar, Dos Hermanas, Seville
  - Virgen del Rocío Hospital, Seville, Seville
  - Hospital Francesc de Borja, Gandia, Valencia